CLINICAL TRIAL: NCT00473915
Title: Intranasal Steroids Prevent Antigen-Induced Hyperresponsiveness of the Nasal Ocular Response
Brief Title: Intranasal Steroids and the Nasal Ocular Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, Professor, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15061B
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone furoate — corticosteroid nasal spray

SUMMARY:
Eye symptoms of tearing, redness and itch frequently occur in patients with allergic rhinitis or hayfever. The purpose of this study is to learn whether placing allergen (the substance that causes allergies) in the nose several days in a row will cause an increase in eye symptoms and whether receiving a nasal steroid spray will prevent these eye symptoms.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 45 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in ocular symptoms | between days 1 and 3

SECONDARY OUTCOMES:
number of eosinophils | between days 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Robert m Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Baroody FM, Shenaq D, DeTineo M, Wang J, Naclerio RM. Fluticasone furoate nasal spray reduces the nasal-ocular reflex: a mechanism for the efficacy of topical steroids in controlling allergic eye symptoms. J Allergy Clin Immunol. 2009 Jun;123(6):1342-8. doi: 10.1016/j.jaci.2009.03.015. Epub 2009 May 9. PMID 19428097